CLINICAL TRIAL: NCT03281837
Title: A Post-market, Single Blind, Multicenter, Randomized, Controlled Trial of HYMOVIS® Intra-articular Injections in Active Subjects With Knee Osteoarthritis
Brief Title: 2 Weekly Intra-articular Hyaluronan Knee Injections, Given 1 wk. Apart, of HYMOVIS Combined With Physical Exercise Program (PEP) Compared to PEP Alone, in Relatively Young, Active Population of Subjects With Patellofemoral Osteoarthritis (PFOA) and/or Tibiofemoral Osteoarthritis (TFOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Pharma USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EQE7-16-01
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis; Patellofemoral Osteoarthritis
Keywords: osteoarthritis; knee osteoarthritis; patellofemoral osteoarthritis; tibiofemoral osteoarthritis; hyaluronan; hyaluronic acid; intra-articular; arthritis; joint disease; active; viscosupplements; Hymovis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Joint Diseases; Motor Activity | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: This post-market, single blind, multicenter, randomized, controlled clinical study is designed to enroll a relatively young, active population of subjects with patellofemoral osteoarthritis (PFOA) and/or tibiofemoral osteoarthritis (TFOA), and to compare responses to treatment with HYMOVIS injections combined with a physical exercise program (PEP) to PEP alone. The study provides for subjects randomized to the PEP alone study group to cross over to HYMOVIS+PEP if improvement has not been achieved by the 3 month follow up visit.
  Subjects will be recruited over a 18 month period. The duration of the trial per center will be approximately 27 months. This includes the enrollment period of 6 months, the follow-up period at 3 and 6 months and the additional follow-up period for patients who crossed-over; they will be followed for an additional 6 months following the initial 3month follow-up. The trial will end when the last subject makes the last visit.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a single-blind study. There will be a blinded evaluator who will not be informed about the intervention (Hymovis + PEP or PEP alone) to which study subjects will be randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1: Hymovis plus Physical Exercise Program (PEP) (Experimental): Intra-articular (IA) Hyaluronan (HA) (Hymovis 24mg/3mL) combined with Physical Exercise program (PEP)
  Interventions: Device: HYMOVIS plus Physical Exercise Program (PEP)
- Group 2: Physical Exercise Program (PEP) alone alone (Other): Specified designed Physical Exercise Program (PEP) not combined with any other intervention
  Interventions: Other: Physical Exercise Program (PEP) alone
- Group 3: Cross-Over group (Other): Patients who were randomized to receive only Physical Exercise Program (PEP) alone and do not respond after 3 months to this intervention will have the opportunity to cross-over to receive 2 intra-articular weekly injections, each injection given 1 week apart, of Hymovis.
  Interventions: Device: HYMOVIS plus Physical Exercise Program (PEP)

INTERVENTIONS:
Device: HYMOVIS plus Physical Exercise Program (PEP) — 1 injection of intra-articular (IA) hyaluronan (HA), Hymovis 24mg/3ml, injection per week for 2 weeks combined with at least 8 weeks of Physical Exercise Program (PEP)
  Arms: Group 1: Hymovis plus Physical Exercise Program (PEP); Group 3: Cross-Over group
Other: Physical Exercise Program (PEP) alone — Physical Exercise Program (PEP) alone for at least 8 weeks
  Arms: Group 2: Physical Exercise Program (PEP) alone alone

SUMMARY:
Knee osteoarthritis (OA) is among the most common causes of musculoskeletal pain and disability. At present, there is no cure for OA. Therefore, the primary aims of therapy are to reduce pain, maintain or improve function and mobility, and prevent or slow the progression of adverse changes to the joint tissues, while keeping potential therapeutic toxicities to a minimum. Current treatment guidelines begin with non-pharmacologic modalities, such as patient education, weight loss, and physical therapy. Several exercise-based therapeutic approaches, such as aerobic exercise programs, range-of-motion exercises, and muscle-strengthening exercises are recommended and have shown clinical benefit in randomized, controlled clinical trials. However, non-pharmacologic approaches frequently provide insufficient pain relief and restoration of function and mobility, and pharmacologic modalities become necessary. Although simple analgesics such as acetaminophen provide relief for many OA subjects with mild to moderate pain, alternatives should be considered for subjects who fail to obtain adequate symptomatic relief with these measures.

This post-market, single blind, multicenter, randomized, controlled clinical study is designed to enroll a relatively young, active population of subjects with patellofemoral osteoarthritis (PFOA) and/or tibiofemoral osteoarthritis (TFOA), and to compare responses to treatment with 2 weekly intra-articular (IA) hyaluronan (HA) injections, with each injection given 1 week apart, of HYMOVIS combined with a physical exercise program (PEP) to PEP alone. Because PEP or exercise programs may be considered the first line standard of care in OA knee pain, particularly in younger, active patients, the hypothesis of the study is that Hymovis combined with PEP program provides greater relief of pain associated with knee OA in the enrolled study subjects than with use of PEP alone.

The study provides for subjects randomized to the PEP alone study group to cross over to HYMOVIS+PEP if improvement has not been achieved by the 3 month follow up visit.

Subjects will be recruited over an 18 month period. The duration of the trial per center will be approximately 27 months. This includes the enrollment period of 6 months, the follow-up period at 3 and 6 months and the additional follow-up period for patients who crossed-over; they will be followed for an additional 6 months following the initial 3month follow-up. The trial will end when the last subject makes the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥21 years and ≤60 years old and with BMI ≤40
* Moderate to severe knee OA pain ≥3 and ≤8 on the NRS pain subscale in the affected knee (signal knee)
* Mild or no pain ≤3 on the numeric rating scale (NRS) pain subscale in the contralateral knee (unaffected knee)
* Persistent knee pain lasting at least 3 months prior to Screening
* Active life-style (play or train themselves at least 2 to 3 times per week)
* Diagnosis of knee OA confirmed by radiographic assessment (must be performed within 6 months prior to screening visit):

  1. anterior-posterior view (weight bearing extension or semi-flexion) of tibiofemoral joint, (posterior-anterior/Rosenberg view as an additional alternate)
  2. lateral view of both the tibiofemoral and patellofemoral joints
  3. Merchant X-ray (or Sunrise) view for patellofemoral joint.
* Radiographic assessment must confirm K-L Grade 1 to 3 for TFOA and/or K-L Grade 1 to for PFOA.
* Radiographic assessment confirms normal articulation of patella and trochlea in Merchant (or Sunrise) view

Exclusion Criteria:

* Radiographic assessment confirms abnormal patellofemoral tracking or articulation in lateral and/or Merchant view (or Sunrise View)
* Major injury to or disorder of the contralateral knee or other weight-bearing joint that would interfere with the study assessments.
* Secondary OA of the study joint due to a prior or concomitant condition (e.g., septic arthritis, inflammatory joint disease, gout, articular fracture, major dysplasia, or congenital abnormality, hemochromatosis, etc.).
* Surgery to the study joint within the previous 12 months prior to Screening. Surgery to the contralateral knee or other weight-bearing joint within the previous 12 months that would interfere with the study assessments.
* Patients with either total joint replacement implants, unicondylar implants or patellofemoral replacement implants in the affected joint.
* Ligament reconstruction of the affected knee within 3 years.
* Inflammatory arthropathies such as rheumatoid arthritis, lupus, or psoriatic arthritis.
* Episode of gout or calcium pyrophosphate (pseudogout) diseases within 6 months prior to Screening.
* IA or local peri-articular corticosteroid injections to the study joint/knee within 8 weeks (2 months) prior to Screening or to any other joint (other than the study joint) or soft tissue area within 1 month prior to Screening.
* Any oral corticosteroid within 1 month prior to Screening. Steroid inhalants are permitted if the Subject has been on a stable regimen for the past 1 month prior to Screening and remains on this regimen throughout the course of the trial.
* Intra-articular HA in the study joint within 6 months prior to Screening.
* History of allergic reaction to an intra-articular Hyaluronic acid injection.
* Known hypersensitivity (allergy) to gram positive bacterial proteins.
* Use of glucosamine or chondroitin sulfate containing products unless the subject is on stable doses for at least 14 days prior to Screening and willing to remain on these stable doses throughout the course of the study.
* Inability to perform the climbing stair test.
* X-ray findings of acute fractures, severe loss of bone density, avascular necrosis and/or severe deformity.
* Axial deviation of the lower limbs greater than 20 degrees in valgus or varus on standing X-ray.
* Symptomatic OA of either hip or spine with a pain score ≥2 on the NRS on or off pain medication.
* Clinically significant medio-lateral and/or anterior-posterior instability.
* Osteonecrosis of either knee.
* Participation in a physical therapy regimen that has not been stable during the 1 month prior to Screening and the subject is unwilling or unable to maintain the same regimen throughout the course of the trial or is unwilling to stop previously prescribed or self-initiated physical therapy regimen and switch solely to and initiate study defined PEP program.
* K-L Grade 4 TFOA of the knee (i.e., large osteophytes, marked narrowing, severe sclerosis, and definite deformity).
* K-L Grade 4 PFOA of the knee (i.e., large osteophytes, marked narrowing, severe sclerosis, definite deformity)
* Hemiparesis of the lower limbs.
* Significant surgery of lower limbs (hip, ankle, foot) that may interfere with knee assessments.
* Chronic use of analgesia for pain (including pain in the other knee or any other joint) that may interfere with the evaluations of the test knee (such as possible use of rescue medication for these other conditions).
* Known allergies to acetaminophen and hyaluronan preparations.
* Know hypersensitivity (allergy) to anesthetics
* Recurrent medical history of severe allergic or immune-mediated reactions.
* Active infection or skin diseases in the area of the potential injection site or joint.
* Any dermatological disease overlying the signal joint that would contraindicate multiple injections or aspirations.
* Use of any agent reported to have symptom relief for arthritis or be a disease/structure modifying drug (e.g. doxycycline, long-term tetracycline, s-adenosylmethionine [SAM], methylsulfonylmethane [MSM] or dimethylsulfoxide [DMSO], dietary supplements or any herbal remedy taken for arthritic and joint conditions within the past month (exceptions as specified in Exclusion #14).
* Peripheral neuropathy that would be severe enough to interfere with the evaluation of the subject.
* Psychological status (e.g., anxiety, depression, poor sleep quality, pain catastrophizing, etc.) that may interfere with functional assessment of the target knee.
* Vascular insufficiency of lower limbs that is severe enough to interfere with the evaluation of the subject.
* Concomitant therapy with anticoagulants (low dose aspirin, not exceeding 325 mg per day as an anti-thrombotic agent is permitted if stable for 1 month prior to Screening and remains stable throughout the study).
* Any concomitant disease(s) or condition(s) that may interfere with the free use and evaluation of the affected knee for the 6 months course of the trial (cancer, other rheumatic diseases, gout, severe congenital defects, etc.).
* Any serious mobility problems (e.g. Parkinson's disease) or claustrophobia
* Any concomitant chronic disease(s) or condition(s) that may predispose them to a high probability of interfering with the completion of the 6-month follow-up of the study such as peptic ulcer, liver disease, severe coronary disease, renal disease, cancer, pregnancy, alcoholism, drug abuse, mental state, or other clinically significant condition.
* Excessive alcohol consumption or alcoholism that would be contraindicated with the use of acetaminophen.
* Use of marijuana, whether prescribed or not
* Any clinically significant diagnostic test and/or abnormal laboratory test result(s) that, in the opinion of the clinical investigator, may place the subject's health at risk, impact the study, or impact the subject's ability to complete the study.
* Inability to legally comprehend the details and nature of the study for any reason, including psychiatric illness.
* Likelihood of protocol violations or unlikely to compete the study for any reason, as determined by the clinical investigator.
* Continued participation in an experimental drug/device study or any clinical trial within the previous 8 weeks prior to Screening. Subjects must have fully completed participation in an experimental drug/device study of any clinical trial at least 8 weeks prior to screening.
* Pregnancy, breastfeeding, planned conception, premenopausal women who have not had tubal ligation, hysterectomy, or are unwilling or unable to utilize contraceptive measures (or contraception)
* Prior history of any malignancy with the exception of basal cell carcinoma of the skin treated more than 2 years prior to Screening.
* Significant bleeding diathesis.
* Participation in current litigation for injuries related to the study knee or other injuries that might interfere with their completion of the study protocol.
* Non-English speaking subjects.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Improvement in average score for 4 of the 5 Knee Injury and Osteoarthritis Outcome Score subscales (KOOS) over 3 months from baseline (Day 90). Scores to be measured are pain, symptoms, function in sport and recreation, and knee related quality of life. | Baseline and 90 days after baseline

SECONDARY OUTCOMES:
Safety - Number of participants with intervention / treatment-related adverse events | Baseline, 30 days, 60 days, 90 days, 120 days, 150 days, 180 days, through study completion (1 year)
  The investigator's determination and term of each adverse event (AE) will be mapped to system organ class and preferred term using the MedDRA dictionary. Incidence and frequency of AE's will be summarized for each treatment group by MedDRA system organ class and preferred term. A subject will only be counted once per system organ class and once per preferred term within a treatment. The summaries will include: All adverse events, All adverse events by severity, All adverse events by relationship to the study device, All adverse device effects, All adverse events leading to discontinuation from study
Time to onset and duration of pain relief at all post-baseline points for the duration of the study | Baseline, 30 days, 60 days, 90 days, 120 days, 150 days, 180 days, through study completion (1 year)
Number of subjects achieving pain-free or disability-free return to sports over the duration of the study | Baseline, 30 days, 60 days, 90 days, 120 days, 150 days, 180 days, through study completion (1 year)
Analysis on the need for rescue analgesic medication for pain relief | Baseline, 30 days, 60 days, 90 days, 120 days, 150 days, 180 days, through study completion (1 year)
Global assessments and SF-12 conducted by the clinicians and self-reported by the subjects | Baseline, 90 days, 180 days, through study completion (1 year)
Number of subjects continuing to cross-over phase of study due to failure to respond adequately to PEP alone | Baseline, 90 days, 180 days, through study completion (1 year)
Biochemical serum biomarker analysis. | Baseline, 90 days, 180 days, through study completion (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Cedars-Sinai Medical Center, Principal Investigator — Cedars-Sinai Medical Center - Department of Orthopaedic Surgery; Kerlan-Jobe Orthopaedic Clinic, Principal Investigator — Kerlan-Jobe Orthopaedic Clinic
Locations (10):
- United States (10):
  - Tucson Orthopaedic Institute Research Center, Tucson, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Kerlan-Jobe Orthopaedic Clinic, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Horizon Clinical Research / Grossmont Orthopaedic Medical Group, San Diego, California
  - Andrews Institute Orthopaedics and Sports Medicine - Andrews Research & Education Foundation, Gulf Breeze, Florida
  - Cartilage Research Foundation, Inc. - OrthoIndy, Greenwood, Indiana
  - New York University - Center for Musculoskeletal Care, New York, New York
  - Hospital for Special Surgery, New York, New York
  - IntegraTrials LLC / OrthoVirginia, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Undecided